CLINICAL TRIAL: NCT06194825
Title: A Phase 3, Randomized Study, With Initial 24-week, Double-Blind and Placebo-Controlled Treatment Phase, Followed by An 80-week Open-label Extension Treatment Phase to Evaluate the Effect of Eplontersen on the Transthyretin Reduction and Long-Term Safety in Chinese Participants With Transthyretin Amyloid Cardiomyopathy (EPIC-ATTR)
Brief Title: EPIC-ATTR: A Study to Evaluate the Effect of Eplontersen on the Transthyretin Reduction and Long-term Safety in Chinese Subjects With Transthyretin Amyloid Cardiomyopathy
Acronym: EPIC-ATTR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D8450C00005
Record Dates: First submitted 2023-12-05; First posted 2024-01-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Transthyretin Amyloid Cardiomyopathy
Keywords: Eplontersen; ATTR-CM
MeSH Terms: interventions — eplontersen

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized in a 3:1 ratio to either eplontersen or placebo in the double-blind treatment phase, followed by the open label treatment phase (participants initially assigned to placebo will switch to eplontersen treatment from Week 24), to evaluate long term safety and tolerability of eplontersen treatment.
Who Masked: Participant, Investigator
Masking Description: The treatment assignment of the 24-week double-blind treatment phase will be kept blinded to sponsor until the end of double-blind treatment phase and kept blinded to participants and investigators until the end of study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Eplontersen (Experimental): Eplontersen by subcutaneous injection once every 4 weeks
  Interventions: Drug: Eplontersen
- placebo (Placebo Comparator): Eplontersen-matching placebo by subcutaneous injection once every 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eplontersen — Eplontersen by subcutaneous injection
  Arms: Eplontersen
Drug: Placebo — Eplontersen-matching placebo by subcutaneous injection
  Arms: placebo

SUMMARY:
The purpose of this study is to investigate the effect of eplontersen compared to placebo on the reduction of serum TTR concentration and long-term safety in Chinese participants with hereditary or wild-type transthyretin amyloid cardiomyopathy.

DETAILED DESCRIPTION:
This is a Phase 3, randomized study, with initial 24-week double-blind and placebo-controlled treatment phase, then followed by an open-label extension treatment phase to evaluate the effect of eplontersen on the TTR reduction and long-term safety in Chinese participants with ATTR-CM. Eligible participants will be randomized in a 3:1 ratio to either eplontersen or placebo for a treatment period of 24 weeks. The double-blind treatment phase will be followed by 80-week open label treatment phase (Participants initially assigned to placebo will switch to eplontersen treatment at 24 weeks), to evaluate long term safety and tolerability of eplontersen treatment. This study will be performed in about 30 to 35 study centres in China mainland.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated) and any authorizations required by local law and be able to comply with all study requirements.
2. 20 to 90 years of age (inclusive).
3. Females: must be non-pregnant and non-lactating and either:

   1. surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy);
   2. post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the post-menopausal range for the laboratory involved);
   3. abstinent* or,
   4. if engaged in sexual relations of child-bearing potential, agree to use 1 highly effective contraceptive method from the time of signing the informed consent form until at least 24 weeks after the last dose of study intervention (eplontersen or placebo).

   Males must be surgically sterile or abstinent*; if engaged in sexual relations with a female of child-bearing potential, the participant must be using an acceptable contraceptive method from the time of signing the informed consent form until at least 24 weeks after the last dose of study intervention.

   A highly effective method of contraception is defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly, such as implants, injectables, hormonal methods etc.

   *Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception.
4. Willing to be genetically tested for mutations in the TTR gene before study intervention administration, if it was not done before.
5. Amyloid deposits in cardiac or non-cardiac tissue confirmed by Congo Red (or equivalent) staining OR technetium scintigraphy (99mTc-3,3-diphosphono-1,2 propanodicarboxylic acid [DPD-Tc], 99m Tc-pyrophosphate [PYP-Tc], or 99mTc-hydroxymethylene-diphosphonate [HMDP-Tc]) with Grade 2 or 3 cardiac uptake in the absence of abnormal light chains ratio, centrally confirmed.
6. End-diastolic interventricular septum thickness of > 12 mm on screening echocardiogram.
7. Medical history of HF secondary to hereditary or wild-type ATTR-CM with at least:

   1. prior hospitalization for HF, which may include hospitalization for arrhythmia or pacemaker/implantable cardioverter defibrillator placement, or
   2. symptoms and signs of volume overload or elevated intracardiac pressure that requires treatment with diuretics other than mineralocorticoid receptor antagonists for clinical stabilization.
8. Screening NT-proBNP ≥ 600 pg/mL(≥ 1200 pg/mL for participants with atrial fibrillation) by central lab.
9. New York Heart Association (NYHA) class I-III.
10. 6-Minute Walk Distance ≥ 100 meters.
11. If on medical treatment for HF on stable dosage regimen for at least 2 weeks prior to randomization.
12. Willing to adhere to vitamin A supplementation per protocol.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Acute coronary syndrome, unstable angina, stroke, TIA, coronary revascularization, cardiac device implantation, cardiac valve repair, or major surgery within 3 months prior or during screening.
2. Hospitalization or urgent visit to emergency department/emergency room for worsening of HF with discharge date within 4 weeks prior to or during screening.
3. Uncontrolled hypertension (systolic BP > 160 mmHg or diastolic BP > 100 mmHg).
4. Uncontrolled clinically significant cardiac arrhythmia, per investigator's assessment (e.g., no pacemaker, although indicated).
5. Severe uncorrected cardiac valvular disease.
6. Cardiomyopathy not primarily caused by ATTR-CM, for example, cardiomyopathy due to hypertension, valvular heart disease, or ischemic heart disease.
7. Screening laboratory results as follows, or any other clinically significant abnormalities in screening laboratory values that would render a participant unsuitable for inclusion, per investigator's assessment.

   1. Alanine aminotransferase/aspartate aminotransferase (ALT/AST) > 2.0 × ULN.
   2. Total bilirubin ≥ 2.0 × ULN (participants with total bilirubin ≥ 2.0 × ULN may be allowed on study if indirect bilirubin only is elevated, ALT/AST is not greater than the ULN and known to have Gilbert's disease OR if, in the opinion of the investigator, the bilirubin abnormality is deemed not clinically significant, pending proper follow-up with the local specialist and discussion with Medical Monitor).
   3. Platelets < 125 × 109/L.
   4. Urine protein creatinine ratio (UPCR) ≥ 750 mg/g. In the event of UPCR above this threshold ineligibility may be confirmed by a repeat random spot UPCR UPCR ≥ 750 mg/g.
   5. Positive test for blood (including trace) on urinalysis that is subsequently confirmed with urine microscopy showing > 5 red blood cells per high power field and is related to glomerulopathies. In women, this exclusion criterion must be assessed outside of menstrual period. If in the opinion of the investigator the hematuria is not considered related to glomerulopathies the participant may be considered eligible, pending proper follow-up and a discussion with the Medical Monitor. Participants with history of bladder cancer must have been treated with curative intent and have not presented recurrence within the prior 5 years.
   6. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 at screening (CKD EPI formula [Levey et al. 2009]). If the eGFR is thought to be underestimated, the CKD EPI creatinine-cystatin C equation can be used for confirmation (Inker et al. 2012).
   7. Abnormal thyroid function tests with clinical significance per investigator's judgement.
   8. Serum retinol level at screening < Lower Limit of Normal (LLN). Unless, after ophthalmologist consultation, the investigator considers the retinol level below LLN not clinical relevant. In this case the participant may be considered to be eligible, pending a discussion with the Medical Monitor. (This criterion does not apply to ATTRv-CM patients with known mutation at the position 84 [e.g., Ile84Ser]).
   9. Hemoglobin A1c (HbA1c) > 9.5%.
8. Monoclonal gammopathy of undetermined significance (MGUS) and/or alterations in immunoglobulin FLC ratio, unless fat, bone marrow, or heart biopsy confirming the absence of light chain and the presence of TTR protein by mass spectrometry or immunoelectron microscopy. For participants with CKD and without presence of monoclonal protein in blood and urine, the acceptable FLC ratio is 0.26 to 2.25. Results different from that may be discussed with local hematologist, investigator and Medical Monitor if the risks associated with the biopsy outweigh the benefits.
9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1.
10. Known history of or positive test for HIV (as evidenced by positive tests for HIV antibody), hepatitis C (as evidenced by positive tests for HCV antibody and HCV RNA) or hepatitis B (as evidenced by a positive test for hepatitis B surface antigen).
11. History of bleeding, diathesis or coagulopathy (e.g., liver cirrhosis, hematologic malignancy, antiphospholipid antibody syndrome, congenital disorders such as hemophilia A, B, and Von Willebrand disease).
12. If receiving oral anticoagulants (except vitamin K antagonists), the dose must have been stable for 4 weeks prior to the first dose of study intervention and regular monitoring must be performed, per clinical practice during the study. If the participant is receiving vitamin K antagonists (e.g., warfarin) INR should be in therapeutic range, as established by the investigator, for 4 weeks prior to the first dose.
13. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin, melanoma in situ, prostate carcinoma grade group 1, breast ductal carcinoma in situ, or carcinoma in situ of the cervix. Participants with a history of other malignancies who have been treated with curative intent and without recurrence within 5 years may also be eligible per investigator's judgment.
14. Prior liver or heart transplant, and/or left ventricular assist device (LVAD) or anticipated liver transplant or LVAD within 1 year after randomization.
15. Karnofsky performance status of ≤ 50%.
16. Known Light chain/Primary Amyloidosis.
17. Known leptomeningeal amyloidosis.
18. Known history of multiple myeloma.
19. Treatment with another investigational drug and/or biological agent within 1 month of screening, or 5 half-lives of investigational agent, whichever is longer.
20. Current or previous treatment with Tegsedi™ (inotersen) or Onpattro™ (patisiran) or other oligonucleotide or RNA therapeutic (including siRNA; does not apply to COVID 19 mRNA vaccinations).
21. Current treatment with diflunisal, doxycycline with or without ursodeoxycholic acid, and/or non-dihydropyridine calcium-channel blocker (e.g., verapamil, diltiazem). Participants receiving any of these agents must respect a wash-out period of 14 days before randomization.
22. Unwillingness or inability to comply with study procedures, including follow-up, as specified by this protocol, or unwillingness to cooperate fully with the investigator. For completing PRO assessments, participants who are unable to read (e.g., are blind or are illiterate) should be excluded from participating in this trial.
23. Other physical, social, or psychological conditions including illicit drug or alcohol use, which, in the opinion of the investigator would make the participant unsuitable for inclusion, or could interfere with the participant participating in or completing the study.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-05-14 (Estimated); Study Completion 2027-01-05 (Estimated)

PRIMARY OUTCOMES:
Percent change of serum TTR concentration from baseline | up to 24 weeks
  To evaluate the effect of eplontersen compared to placebo on serum transthyretin (TTR) concentration up to 24 weeks

SECONDARY OUTCOMES:
Changes from baseline in NT-proBNP serum level | up to 24 weeks
  To evaluate the effect of eplontersen compared to placebo up to 24 weeks in NT-proBNP serum level
Changes from baseline in hs-cTnT serum level | up to 24 weeks
  To evaluate the effect of eplontersen compared to placebo up to 24 weeks in hs-cTnT serum level
Plasma concentrations of eplontersen at specified time-points (Week0,2,4,8,12,16,20,24,28,32,36,48,60,72,84,96,104) | up to 124 weeks
  To evaluate the pharmacokinetics (Ctrough) of eplontersen
Plasma concentrations of anti-drug antibodies (ADA) at specified time-points (Week0,2,4,8,12,16,20,24,28,32,36,48,60,72,84,96,104,114,124) | up to 124 weeks
  Including but not limited to anti-drug antibodies (ADA) prevalence and incidence, different ADA status (treatment induced, treatment-boosted and treatment-unaffected ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Shuyang Zhang, MD, Principal Investigator — Peking Union Medical College
Locations (14):
- China (14):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Ha’erbin
  - Research Site, Jinan
  - Research Site, Nanchang
  - Research Site, Shanghai
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Wuhan
  - Research Site, Xi'an